CLINICAL TRIAL: NCT07179874
Title: Effects of Remote Ischemic Preconditioning on Contrast-Induced Kidney Damage in Diabetic Patients: Link to Oxidative Stress
Brief Title: Remote Ischemic Preconditioning to Prevent Contrast-Induced Kidney Injury in Diabetic Patients (PRINCES)
Acronym: PRINCES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Collaborators: Hospital General Universitario Santa Lucía (Other)
Responsible Party: Principal Investigator, Francisca Rodriguez Mulero, Associate Professor, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Tl14-13 MGM
Record Dates: First submitted 2025-08-15; First posted 2025-09-18 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Contrast-induced Acute Kidney Injury
Keywords: Remote Ischemic Preconditioning; Diabetes Mellitus; Heme Oxygenase-1
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Participants were randomized using block randomization with sealed opaque envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote ischemyc preconditioning. (Experimental): Participants assigned to this arm received:
  * Standard hydration therapy: intravenous infusion of 0.9% saline at 1 ml/kg/h for 12 hours before and after coronary catheterization
  * Plus the RIPC procedure: four alternating cycles of upper-arm ischemia (inflating a blood pressure cuff 50 mmHg above systolic pressure for 5 minutes, followed by 5 minutes of reperfusion) performed approximately 45 minutes before catheterization This group was intended to assess the protective renal effects of RIPC in diabetic patients undergoing exposure to intravenous contrast media.
  Interventions: Procedure: Remote Ischemic Preconditioning
- Control Arm-NO RIPC (No Intervention): Participants in the control arm receive standard care without remote ischemic preconditioning (RIPC). All patients undergo intravenous hydration as part of standard preventive measures prior to coronary catheterization.
  * Intervention: 0.9% saline solution administered intravenously at a rate of 1 ml/kg/hour
  * Timing: Initiated 12 hours before the procedure and maintained for 12 hours afterward
  * Additional Notes: No cuff inflation or ischemic maneuvers are performed. Patients do not receive sham stimulation or any form of simulated ischemia. This arm reflects usual clinical practice in patients undergoing catheterization who meet inclusion criteria.

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning — This intervention involves a non-invasive, mechanical stimulus applied to an upper limb with the goal of activating systemic protective pathways against contrast-induced nephropathy in diabetic patients. Unlike pharmacologic or device-based interventions, RIPC:
  * Does not involve any drugs, biologics, or implants
  * Is performed using a standard blood pressure cuff, inflated to 50 mmHg above systolic pressure, specifically designed to induce repetitive transient limb ischemia
  * Consists of four alternating cycles of 5 minutes inflation followed by 5 minutes reperfusion
  * Is applied 45 minutes before coronary catheterization, timed to optimize systemic renal protection prior to exposure to contrast media
  * Targets activation of the heme oxygenase-1 (HO-1) enzymatic pathway, linking limb ischemia with antioxidant renal defense mechanisms Unlike interventions that rely solely on hydration or pharmacological antioxidants, this approach seeks to prime endogenous protective systems through is
  Arms: Remote ischemyc preconditioning.

SUMMARY:
This study investigates whether remote ischemic preconditioning (RIPC)-a non-invasive technique involving brief cycles of blood flow restriction to the arm-can prevent contrast-induced nephropathy (CIN) in diabetic patients undergoing coronary angiography. Diabetes mellitus increases the risk of CIN due to heightened oxidative stress and disrupted protective cellular signaling.

While previous research suggests that RIPC may activate renal protective mechanisms, its efficacy in diabetic individuals remains controversial, as metabolic and neurovascular alterations may compromise its effect. This randomized trial aims to determine whether RIPC reduces oxidative kidney damage and improves renal outcomes in this high-risk population. The study will also explore the biological basis for potential variability in response, focusing on oxidative stress biomarkers and early kidney injury indicators.

DETAILED DESCRIPTION:
This clinical trial explores a non-invasive method known as Remote Ischemic Preconditioning (RIPC) to prevent contrast-induced kidney damage in people with diabetes who are undergoing coronary catheterization. RIPC involves applying brief cycles of restricted blood flow to the arm using a pressure cuff before a medical procedure. Research suggests that RIPC may trigger protective biological responses in distant organs, such as the kidneys, by activating endogenous defense mechanisms including the antioxidant enzyme heme oxygenase-1 (HO-1), and modulation of inflammatory pathways.

The study focuses on a serious complication called Contrast-Induced Nephropathy (CIN)-an acute kidney injury that can occur in patients exposed to contrast dye during medical imaging. CIN is particularly common and severe among individuals with diabetes mellitus and impaired renal function. In this population, the incidence of CIN may reach up to 90%, leading to adverse clinical outcomes and increased healthcare costs.

One major mechanism implicated in CIN is oxidative stress, a state in which excess reactive oxygen species (ROS) overwhelm the body's antioxidant defenses. This imbalance is even more pronounced in diabetic kidneys, where chronic metabolic dysregulation and endothelial dysfunction contribute to heightened susceptibility.

Although early evidence pointed toward a protective role of RIPC against CIN, growing data suggest that its efficacy may be compromised in diabetic individuals. Diabetes-related impairments-including disrupted intracellular signaling, reduced humoral mediator release, autonomic dysfunction, and increased oxidative stress-could attenuate the protective cascade activated by RIPC. Furthermore, peripheral neuropathy, a common complication affecting up to 50% of diabetic patients, may interfere with the neural transmission necessary for systemic RIPC effects.

Nonetheless, clinical studies such as the RenPro Trial have reported preserved RIPC-mediated protection in diabetic populations undergoing contrast exposure. These divergent findings raise important questions about patient-specific factors-including glycemic control, pharmacotherapy, and comorbid conditions-that may modulate the efficacy of this intervention.

The present study was initially designed to evaluate the protective potential of RIPC in the diabetic population. However, from its inception, the trial also considered the hypothesis that protective mechanisms may be altered or suppressed in diabetes. As such, it aims not only to assess clinical outcomes, but also to explore biological indicators that might explain variability in response.

This randomized, parallel-group trial will be conducted in the intensive care unit (ICU) at Hospital General Universitario Santa Lucía. Participants will include adults with diabetes admitted for acute coronary syndrome and scheduled for coronary angiography. Subjects will be randomly assigned to:

* RIPC + hydration group
* Hydration-only control group All participants will receive standard intravenous fluid therapy before and after contrast administration. Those in the RIPC group will undergo four cycles of cuff-induced limb ischemia and reperfusion immediately prior to the procedure.

Biological samples (blood and urine) will be collected at baseline, 24h, 48h, and 72h after contrast exposure to evaluate:

* Traditional kidney function markers: serum creatinine
* Early kidney injury biomarkers: cystatin C.
* Oxidative stress markers: MDA, HO-1 (plasma, urine, and intracellular)

Secondary outcomes include:

* Duration of ICU and hospital stay
* In-hospital mortality
* Correlation between biomarker profiles and prognosis Laboratory analyses will include ELISA and Western blot techniques, while statistical modeling will assess predictive factors and treatment effects.

This study aims to clarify whether RIPC can offer a reproducible, low-cost strategy to prevent CIN in a high-risk diabetic population, and to deepen understanding of the cellular and systemic mechanisms underpinning renal protection under metabolic stress.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with diabetes mellitus.
* Age above 18 years.
* Admission to the ICU due to acute coronary syndrome.
* Indication for undergoing a coronary arteriography (either urgent or scheduled)
* Patients who received a coronary arteriography within the last 72 hours (if previously recruited, counted as new for randomization).
* Possibility to perform the RIPC maneuver without delaying the catheterization

Exclusion Criteria:

* Absence of diabetes mellitus.
* Pregnant women.
* Renal transplant recipients.
* Patients who underwent urological procedures or received intravenous contrast within the last 72 hours.
* Diagnosis of end-stage renal disease requiring hemodialysis.
* Participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-02-25 (Actual); Primary Completion 2017-01-09 (Actual); Study Completion 2017-01-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Contrast-Induced Nephropathy (CIN), defined as an increase in serum creatinine ≥25% or ≥0.5 mg/dL from baseline within 72 hours after contrast exposure | Time Frame: 24, 48, and 72 hours post-contrast administration
  * Metric: Absolute change in serum creatinine level (mg/dL)
  * Time Frame: 24, 48, and 72 hours post-contrast administration
  * Purpose: Evaluates the incidence and severity of contrast-induced nephropathy (CIN)
  * Rationale: Creatinine is a key biomarker for acute kidney injury, particularly relevant in diabetic populations receiving iodinated contrast agents

SECONDARY OUTCOMES:
- Changes in Heme Oxygenase-1 (HO-1) concentration in plasma . | 24, 48, and 72 hours after contrast administration
  Quantitative change in plasma levels of Heme Oxygenase-1 (HO-1) measured in nanograms per milliliter (ng/mL) using ELISA (ADI-960-071; commercial distributor: Enzo Diagnostics) before and after remote ischemic preconditioning (RIPC).
Duration of ICU/Hospital Stay. | Up to 30 days post-ICU admission
  Total number of days spent in the ICU and hospital.
Survival . | 6 weeks post-hospital discharge
  Survival will be assessed as all-cause mortality.
Hospital Readmission Rate | 6 weeks post-hospital discharge
  Number of patients readmitted to the hospital within 6 weeks post-hospital discharge.
Clinical Status | 6 weeks post-hospital discharge
  Assessment of the patient's clinical condition at discharge (e.g., stable, improved, deteriorated).
Need for Dialysis | 6 weeks post-hospital discharge
  Number of patients requiring renal replacement therapy .

OTHER OUTCOMES:
Neutrophil and Lymphocyte Counts and Neutrophil-to-Lymphocyte Ratio (NLR) | From baseline to 72 hours after coronary catheterization
  Quantitative changes in total neutrophil count, total lymphocyte count, and the derived neutrophil-to-lymphocyte ratio (NLR) calculated from these values in peripheral blood samples collected before and after remote ischemic preconditioning (RIPC).
NT-proBNP Levels (Cardiac Stress Marker) | From baseline to 72 hours after coronary catheterization
  Quantitative change in plasma levels of N-terminal pro-B-type natriuretic peptide (NT-proBNP), measured before and after remote ischemic preconditioning (RIPC) . This marker reflects cardiac stress and was assessed as part of the biochemical profile.
Ferritin (Ft) Levels | From baseline to 72 hours after coronary catheterization
  Quantitative change in plasma ferritin (Ft) levels measured in nanograms per milliliter (ng/mL) before and after remote ischemic preconditioning (RIPC).
C-Reactive Protein (CRP) Levels | From baseline to 72 hours after coronary catheterization
  Quantitative change in plasma C-reactive protein (CRP) levels measured in milligrams per deciliter (mg/dL), before and after remote ischemic preconditioning (RIPC).

CONTACTS AND LOCATIONS:
Overall Officials: FRANCISCA RODRIGUEZ, Ph.D, Principal Investigator — University of Murcia-MURCIA; MARIA DOLORES RODRIGUEZ, M.D. Ph.D., Principal Investigator — Hospital Santa Lucía-CARTAGENA, MURCIA; MARIA GALINDO MARTINEZ, M.D. Ph.D., Principal Investigator — Hospital Santa Lucía-CARTAGENA, MURCIA

IPD SHARING:
Plan to Share IPD: Yes
Description: Individual participant data (IPD) and related data dictionaries will be made available to qualified researchers upon reasonable request. The data sharing will be subject to restrictions, including the requirement for prior approval by all principal investigators involved in the study. Access will be granted only after review of the research proposal to ensure it aligns with ethical and scientific standards.
  Time Frame: Beginning 6 months after publication of the primary results; data available for up to 2 years.
  Access Criteria: Researchers must submit a detailed, methodologically sound proposal and sign a data use agreement that protects participant confidentiality.
  Access Mechanism: Data will be shared through a secure institutional repository or directly by the study sponsor upon approval.
Supporting Information: CSR
Time Frame: Beginning 6 months after publication of the primary results; data available for up to 2 years.
Access Criteria: Researchers must submit a detailed, methodologically sound proposal and sign a data use agreement that protects participant confidentiality

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT07179874/Prot_SAP_000.pdf
  • Informed Consent Form (2025-09-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT07179874/ICF_001.pdf